CLINICAL TRIAL: NCT00870116
Title: SBRT Radiotherapy for Non-operated Non-small-cell Lung Cancer (NSCLC), T1-T2, N0, M0
Brief Title: Stereotactic Body Radio Therapy (SBRT) for Early-stage Non Small Cell Lung Cancer (NSCLC)
Acronym: SBRT-NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: The Biostatistics and Therapy Evaluation Unit (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBRT CNPC; ET2008-067
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: SBRT; non-operated; non-metastatic; non-small-cell lung cancer; conformational radiotherapy; non-operated non-metastatic non-small-cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - SBRT using cyberknife (Other): SBRT using cyberknife: treatment = 2x15 Gy during 2 weeks
  Interventions: Radiation: SBRT by cyberknife
- 2 - SBRT using linear accelerator (Other): SBRT using linear accelerator: treatment = 2x15 Gy during 2 weeks
  Interventions: Radiation: SBRT by linear accelerator
- 3 - Conformational radiotherapy (Other): Conformational radiotherapy: treatment = 5x2 Gy during 7 weeks
  Interventions: Radiation: Conformational radiotherapy

INTERVENTIONS:
Radiation: SBRT by cyberknife — treatment = 2x15 Gy during 2 weeks
  Arms: 1 - SBRT using cyberknife
Radiation: SBRT by linear accelerator — treatment = 2x15 Gy during 2 weeks
  Arms: 2 - SBRT using linear accelerator
Radiation: Conformational radiotherapy — treatment = 5x2 Gy during 7 weeks (free breathing or breath holding)
  Arms: 3 - Conformational radiotherapy

SUMMARY:
The purpose of this study is to evaluate local disease control after 2 years in patients with non-metastatic, non-operated non-small-cell lung cancer treated by radiotherapy.

Eligible patients will be recruited and registered consecutively (no randomization). The estimated inclusion period is approximately 24 months. The duration of the research is 4 years.

The number of patients required in this multicentric prospective study is 120:

* 20 patients in the SBRT-1 arm (cyberknife),
* 80 patients in the SBRT-2 arm (linear accelerator-based)
* 20 patients in the conformational radiotherapy arm.

This is a prospective, multicentric, non comparative and non randomized study.

DETAILED DESCRIPTION:
The main objective of this study is to do a health economic evaluation of innovating techniques in radiotherapy.

SBRT is the very precise delivery of high-powered radiation to small target volumes, using multiple low-intensity beams. Extremely precise patient positioning and target location is essential for accurate treatment delivery.

Several studies have shown a benefit of SBRT in terms of local control and progression-free survival, in particular for the treatment of cerebral metastases of limited number and size.

The development of this technique is recent. The number of treatment sessions is low: 1 to 4.

But the patient is exposed to a major risk of toxicity in several organs: the bronchi, the lungs, large vessels, the oesophagus and the spinal-cord.

Pulmonary SBRT imposes strict rules and the use of specific equipment.

Extra-cranial SBRT can be realized using either:

* Conventional linear-accelerator equipped SBRT,
* Cyberknife SBRT.

  3 groups of treatment will be evaluated in this study:
* SBRT by cyberknife,
* SBRT by linear accelerator,
* Conformational radiotherapy (free breathing or breath holding).

ELIGIBILITY:
Inclusion Criteria:

* Non-operated non-small-cell lung cancer (NSCLC) (inoperable tumor or patient refusal of surgery)

  * cytologically or histologically proven NSCLC Or
  * primitive pulmonary tumor of unproven malignancy
* macroscopically normal bronchial endoscopy, negative cytology and biopsies
* AND size increase on 2 successive scans (at 10-12 weeks interval)
* AND hypermetabolic PET-CT pattern
* AND absence of other proven etiology
* Tumor < 5cm, distant (> 1.5 cm) from large vessels, principally in the bronchus and spinal-cord
* No metastasis: M0
* No lymph node involvement: N0
* Functional respiratory evaluation (FRE) compatible with thoracic irradiation
* Maximum expiratory flow-volume > 30% theoretical value
* Age >= 18
* ECOG PS <= 2
* Female patients of childbearing potential: effective method of contraception
* Written advice of the RCP (conciliation meeting) present in the patient file
* Mandatory affiliation with a social security system
* Written, signed informed consent

Exclusion Criteria:

* Previously operated tumors
* Previous thoracic irradiation
* Previous or concurrent primary malignancies at other sites (except basocellular skin cancer or cervical cancer in situ or complete remission for more than 5 years)
* Life expectancy < 6 months
* Pregnant or lactating woman
* Difficult follow-up
* Patient deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of local control in patients with non-operated, non-metastatic non-small-cell lung cancer treated by radiotherapy | 2 years

SECONDARY OUTCOMES:
Health economic evaluation of the various methods used for stereotactic radiotherapy | during treatment / post treatment
Prospective evaluation of acute and late toxicities of SBRT | M1, M3, M6, M12, M18 and M24
Study of quality of life in the 3 groups | inclusion, M1, M3, M12
Evaluation of progression-free survival and overall survival in the 3 groups | No time

CONTACTS AND LOCATIONS:
Overall Officials: Line CLAUDE, MD, Principal Investigator — Centre Léon Bérard, Lyon
Locations (9):
- France (9):
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Val d'Aurelle Paul Lamarque, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Tenon, Paris
  - CHLS, Pierre-Bénite
  - Centre René Gauducheau, Saint-Herblain
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Noel G, Bollet MA, Noel S, Feuvret L, Boisserie G, Tep B, Delattre JY, Baillet F, Ambroise Valery C, Cornu P, Mazeron JJ. Linac stereotactic radiosurgery: an effective and safe treatment for elderly patients with brain metastases. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1555-61. doi: 10.1016/j.ijrobp.2005.04.037. Epub 2005 Jul 18. PMID 16024180
- [Background] Kaplan EL., MP. Nonparametric estimation from incomplete observations. 1958. J Am Stat Assoc 1958; 53:457-481
- [Background] Pommier P. Modélisation spatiale et médico-économique des thérapeutiques innovantes : à propos du projet français ETOILE d'hadronthérapie par ions carbone. Thèse de Science en économie de la santé ; juin 2005
- [Background] Pommier P, Ndiaga Gueye N, Buron C, Meyroneinc S. Modélisation du coût de l'innovation thérapeutique pour l'aide à la décision. Application à la radiothérapie par ions carbone (projet ETOILE). Santé et systémique 2007 ; 10 : 217-31
- [Result] Evaluation de la radiothérapie fractionnée en condition stéréotaxiques des métastases cérébrales, STIC 2005
- [Result] Tschung Sibley G. Radiotherapy for patient with medically inoperable stage I non-small cell lung cancer smaller doses and higher doses - a review. Cancer 2003;41:1-11
- [Result] Timmerman R, Papiez L, McGarry R, Likes L, DesRosiers C, Frost S, Williams M. Extracranial stereotactic radioablation: results of a phase I study in medically inoperable stage I non-small cell lung cancer. Chest. 2003 Nov;124(5):1946-55. doi: 10.1378/chest.124.5.1946. PMID 14605072
- [Result] McGarry RC, Papiez L, Williams M, Whitford T, Timmerman RD. Stereotactic body radiation therapy of early-stage non-small-cell lung carcinoma: phase I study. Int J Radiat Oncol Biol Phys. 2005 Nov 15;63(4):1010-5. doi: 10.1016/j.ijrobp.2005.03.073. Epub 2005 Aug 22. PMID 16115740
- [Result] Whyte RI, Crownover R, Murphy MJ, Martin DP, Rice TW, DeCamp MM Jr, Rodebaugh R, Weinhous MS, Le QT. Stereotactic radiosurgery for lung tumors: preliminary report of a phase I trial. Ann Thorac Surg. 2003 Apr;75(4):1097-101. doi: 10.1016/s0003-4975(02)04681-7. PMID 12683544
- [Result] Xia T, Li H, Sun Q, Wang Y, Fan N, Yu Y, Li P, Chang JY. Promising clinical outcome of stereotactic body radiation therapy for patients with inoperable Stage I/II non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):117-25. doi: 10.1016/j.ijrobp.2006.04.013. Epub 2006 Jun 9. PMID 16765528
- [Result] Nagata Y, Takayama K, Matsuo Y, Norihisa Y, Mizowaki T, Sakamoto T, Sakamoto M, Mitsumori M, Shibuya K, Araki N, Yano S, Hiraoka M. Clinical outcomes of a phase I/II study of 48 Gy of stereotactic body radiotherapy in 4 fractions for primary lung cancer using a stereotactic body frame. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1427-31. doi: 10.1016/j.ijrobp.2005.05.034. Epub 2005 Sep 19. PMID 16169670
- [Result] Onishi H, Araki T, Shirato H, Nagata Y, Hiraoka M, Gomi K, Yamashita T, Niibe Y, Karasawa K, Hayakawa K, Takai Y, Kimura T, Hirokawa Y, Takeda A, Ouchi A, Hareyama M, Kokubo M, Hara R, Itami J, Yamada K. Stereotactic hypofractionated high-dose irradiation for stage I nonsmall cell lung carcinoma: clinical outcomes in 245 subjects in a Japanese multiinstitutional study. Cancer. 2004 Oct 1;101(7):1623-31. doi: 10.1002/cncr.20539. PMID 15378503
- [Result] Hof H, Herfarth KK, Munter M, Hoess A, Motsch J, Wannenmacher M, Debus J J. Stereotactic single-dose radiotherapy of stage I non-small-cell lung cancer (NSCLC). Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):335-41. doi: 10.1016/s0360-3016(02)04504-2. PMID 12738306
- [Result] Uematsu M, Shioda A, Suda A, Fukui T, Ozeki Y, Hama Y, Wong JR, Kusano S. Computed tomography-guided frameless stereotactic radiotherapy for stage I non-small cell lung cancer: a 5-year experience. Int J Radiat Oncol Biol Phys. 2001 Nov 1;51(3):666-70. doi: 10.1016/s0360-3016(01)01703-5. PMID 11597807
- [Result] Fukumoto S, Shirato H, Shimzu S, Ogura S, Onimaru R, Kitamura K, Yamazaki K, Miyasaka K, Nishimura M, Dosaka-Akita H. Small-volume image-guided radiotherapy using hypofractionated, coplanar, and noncoplanar multiple fields for patients with inoperable Stage I nonsmall cell lung carcinomas. Cancer. 2002 Oct 1;95(7):1546-53. doi: 10.1002/cncr.10853. PMID 12237924
- [Result] Lax I, Blomgren H, Naslund I, Svanstrom R. Stereotactic radiotherapy of malignancies in the abdomen. Methodological aspects. Acta Oncol. 1994;33(6):677-83. doi: 10.3109/02841869409121782. PMID 7946448
- [Result] Blomgren H, Lax I, Naslund I, Svanstrom R. Stereotactic high dose fraction radiation therapy of extracranial tumors using an accelerator. Clinical experience of the first thirty-one patients. Acta Oncol. 1995;34(6):861-70. doi: 10.3109/02841869509127197. PMID 7576756
- [Result] Schemper M, Smith TL. A note on quantifying follow-up in studies of failure time. Control Clin Trials. 1996 Aug;17(4):343-6. doi: 10.1016/0197-2456(96)00075-x. No abstract available. PMID 8889347
- [Result] Krol AD, Aussems P, Noordijk EM, Hermans J, Leer JW. Local irradiation alone for peripheral stage I lung cancer: could we omit the elective regional nodal irradiation? Int J Radiat Oncol Biol Phys. 1996 Jan 15;34(2):297-302. doi: 10.1016/0360-3016(95)00227-8. PMID 8567329
- [Result] Gauden SJ, Tripcony L. The curative treatment by radiation therapy alone of Stage I non-small cell lung cancer in a geriatric population. Lung Cancer. 2001 Apr;32(1):71-9. doi: 10.1016/s0169-5002(00)00199-9. PMID 11282431
- [Result] Morita K, Fuwa N, Suzuki Y, Nishio M, Sakai K, Tamaki Y, Niibe H, Chujo M, Wada S, Sugawara T, Kita M. Radical radiotherapy for medically inoperable non-small cell lung cancer in clinical stage I: a retrospective analysis of 149 patients. Radiother Oncol. 1997 Jan;42(1):31-6. doi: 10.1016/s0167-8140(96)01828-2. PMID 9132823
- [Result] Sirzen F, Kjellen E, Sorenson S, Cavallin-Stahl E. A systematic overview of radiation therapy effects in non-small cell lung cancer. Acta Oncol. 2003;42(5-6):493-515. doi: 10.1080/02841860310014453. PMID 14596509
- [Result] Bradley JD, Wahab S, Lockett MA, Perez CA, Purdy JA. Elective nodal failures are uncommon in medically inoperable patients with Stage I non-small-cell lung carcinoma treated with limited radiotherapy fields. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):342-7. doi: 10.1016/s0360-3016(02)04614-x. PMID 12738307